CLINICAL TRIAL: NCT03928275
Title: The Response to Intralesional IL-2 and/or BCG Treatment for Cutaneous Metastatic Melanoma
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Withdrawn prematurely.
Sponsor: Carman Giacomantonio (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Carman Giacomantonio, Surgical Oncologist/General Surgeon/Professor, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 14549
Record Dates: First submitted 2019-04-11; First posted 2019-04-26 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Cutaneous Metastatic Melanoma
Keywords: Interleukin-2; Bacillus Calmette Guerin
MeSH Terms: interventions — Interleukin-2; aldesleukin; BCG Vaccine

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to first stage treatment and allocated to 1) IL-2 or 2) IL-2/BCG treatment. First stage treatment patients receive 4 treatments of 1) IL-2 or 2) IL-2 and BCG. Patient response will be determined for treatment groups following iRECIST guidelines as; 1) complete responder, 2) partial responder, or 3) stable disease. In second stage treatment, patients who completely respond to first stage treatment will be randomized to 1) discontinue treatment and followed every 3 mos for 2 yrs and then every 6 mos from yrs 3-5, or 2) will receive 2 additional treatments and then followed every 3 mos for 2 yrs and then every 6 mos from yrs 3-5. Patients that do not completely respond to first stage treatment, will be re-staged using a PET/CT scan. Patients not requiring escalation to systemic therapy will be randomized and advance to second stage treatment (IL-2, IL-2 and BCG, or BCG).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intralesional IL-2 Treatment (Experimental): CMM patients will received 4 treatments of intralesional Interleukin-2 two weeks apart over an eight week period.
  Interventions: Biological: Interleukin-2
- Combination therapy: Intralesional IL-2 and BCG Treatment (Experimental): CMM patients will receive 4 treatments of combination therapy intralesional Interleukin-2 and Bacillus Calmette Guerin two weeks apart over an eight week period.
  Interventions: Biological: Combination therapy Interleukin-2 and Bacillus Calmette Guerin

INTERVENTIONS:
Biological: Interleukin-2 — IL-2 is prepared as 4 million International Units (IU) per 0.8ml at a total dose of 500,000 IU in 0.1ml of sterilized saline (0.9%, m/v)/lesion.
  Other Names: Proleukin (Aldesleukin)
  Arms: Intralesional IL-2 Treatment
Biological: Combination therapy Interleukin-2 and Bacillus Calmette Guerin — BCG (OncoTICE solutions 1-8 x 10-8 Colony Forming Units (CFU)) will be administered at a maximum dose of 3.2 million CFU per treatment at a maximum of 1.6 million CFU per lesion (max 2 lesions).
  IL-2 is prepared as 4 million International Units (IU) per 0.8ml at a total dose of 500,000 IU in 0.1ml of sterilized saline (0.9%, m/v)/lesion (in remaining lesions).
  Other Names: BCG, strain TICE (OncoTICE) and Proleukin (Aldesleukin)
  Arms: Combination therapy: Intralesional IL-2 and BCG Treatment

SUMMARY:
The investigators aim to include 100 local participants over the next 5 years in a two-stage sequential randomized interventional study of intralesional Interleukin-2 (IL-2) and Bacillus Calmette Guerin (BCG) to assess the utility of treating cutaneous metastatic melanoma (CMM).

DETAILED DESCRIPTION:
In the first stage of the study, all consenting CMM patients will be randomized and will receive 4 treatments of either intralesional IL-2 or intralesional IL-2 and BCG. We hypothesize that patients with MM (stage 3C or 4a with a minimum of 4 lesions) that receive combination therapy (IL-2/BCG) in the first stage of treatment will have a higher complete response (iCR) rate compared to IL-2 therapy alone.

Response to stage-one treatment will be monitored and patient response to treatment will be determined and reported according to Immune Response Evaluation Criteria in Solid Tumours (iRECIST) guidelines. Based on response to stage-one treatment, patients will be placed into a response group before entering stage two. For stage two of the trial, patients will be randomized again, and placed into a treatment group; Il-2, IL-2 and BCG, BCG, or Discontinue Treatment. Response to treatment will be monitored and patient response to treatment will be determined and reported according to iRECIST guidelines.

All patients will have lesions biopsied following standard surgical practice techniques and will provide urine and blood for analysis. Tissue samples will be assessed for immune system activity and transcriptome analysis, and urine and blood will be assessed for immune cell populations and markers. All patients will be followed for 5 years post treatment, and patient disease and survival status will be recorded according to iRECIST.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cutaneous metastatic melanoma.
* Has 4 or more melanoma lesions.
* Between18 and 80 years of age.

Exclusion Criteria:

* Immunocompromized.
* Receiving immuno-therapy for other diagnosis.
* Inflammatory disease.
* Autoimmune disease.
* Pregnant
* HIV
* Test positive for TB

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Number of CMM participants that respond to IL-2 compared to the number of participants that respond to IL-2 and BCG. | 5 years
  The primary outcome measure is the achievement of a superior response rate in patients receiving combination IL-2/BCG treatment compared to patients receiving IL-2 alone. Patient response to treatment will be monitored and patients will be categorized as 1) complete responders, 2) partial responders or 3) stable disease. Data will be analyzed by one-way ANOVA to compare proportion outcomes amongst treatment and response groups.

SECONDARY OUTCOMES:
Number of patients that respond to the addition of BCG in stage two compared to the number of patients respond to continued IL-2 treatment. | 5 years
  The achievement of a superior response rate in patients that partially respond or do not respond to single agent IL-2 in stage one, with the addition of BCG treatment in stage two. Patient response to treatment will be monitored and patients will be categorized as 1) complete responders, 2) partial responders or 3) stable disease. Data will be analyzed by one-way ANOVA to compare proportion outcomes amongst treatment and response groups.
Assessment of overall survival in stage one treatment | 5 years
  Complete responders to stage-one treatments will be assessed to determine if there is a difference in overall survival between participants that continue treatment compared to participants that discontinue treatment. Data will be assessed using Kaplan-Meier methods and compared using Log-rank tests.
Assessment of overall survival in stage two treatment | 5 years
  Response groups following stage-two treatments will be assessed to determine if there is a difference in overall survival amongst response groups. Data will be assessed using Kaplan-Meier methods and compared using Log-rank tests.
Assessment of Disease Progression Within Stage of Disease: Number of stable and/or new metastasis | 5 years
  All patients will be followed every 3 months for 2 years and then biannual assessments for years 3-5 after the initial intervention to assess the number of stable or new lesions amongst treatment response groups. Number (integer value) of new metastases will be recorded as a part of this assessment. Data will be compared using a one-way ANOVA. Post-Hoc analysis will be conducted when needed.
Assessment of Metastasis | 5 years
  Assessment of Metastasis - All patients will be followed every 3 months for 2 years and then biannual assessments for years 3-5 after the initial intervention to assess change in lesion size according to iRECIST guidelines. Lesions will be measured in mm in 2 dimensions as part of this assessment. Data will be compared using a one-way ANOVA. Post-Hoc analysis will be conducted when needed.

CONTACTS AND LOCATIONS:
Overall Officials: Carman A Giacomantonio, MD, Principal Investigator — Nova Scotia Health Authority

IPD SHARING:
Plan to Share IPD: No